CLINICAL TRIAL: NCT06911190
Title: Ten Year Follow-up in FSHD; the FOCUS-3 Study
Brief Title: Ten Year Follow-up in FSHD: the FOCUS 3 Study
Acronym: FSHD-FOCUS 3
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: FSHD-FOCUS 3
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: FSHD - Facioscapulohumeral Muscular Dystrophy
Keywords: FSHD; facioscapulohumeral muscular dystrophy; FSHD1; FSHD2
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FOCUS 3 cohort: Genetically proven FSHD patients

SUMMARY:
This study aims to assess longitudinal data in 170 adult and 30 pediatric genetically and clinically well-defined facioscapulohumeral dystrophy (FSHD) patients. FSHD is a chronic progressive disorder associated with major disability due to loss of function and independence. The clinical variability of FSHD is partially explained by currently known (epi)genetic factors. Identifying the variables that influence the clinical variability is essential for developing targeted therapies. Furthermore, it is crucial to assess the natural course, determine sensitive outcome measures and biomarkers to prepare for future trials. Objective This is a longitudinal study on 200 Dutch FSHD patients with a follow-up of ten years. We will hereby assess the natural disease course; determine the sensitivity to change of clinical outcome measures and muscle imaging; validate newly developed outcome measures; and help identify biomarkers and modulators of disease severity.

Study population: Genetically proven FSHD patients: All 162 patients that participated in the FSHD-FOCUS study, together with all 18 pediatric patients that participated in the iFocus study , and additional 65 newly included patients. Main study parameters/endpoints: Natural history will be assessed by 'traditional' clinical outcome measures: Motor Function Measure D1, Ricci-score, MRC scores and FSHD clinical score for adults. Additionally in children shoulder dysfunction performance of upper limb and Facial weakness score will be assessed. Natural history will also be quantified using newer clinical outcome measures and patient-reported measures: Reachable workspace, FSHD-RODS and FSHD Facial Function scale in adults. In children, Reachable workspace and FSHD-COM Peds will be assessed. Muscle MRI and ultrasound will be performed to determine progression of fat replacement, fibrosis, and muscle inflammation.

Furthermore, blood samples will be taken in adult participants for (epi)genetic analysis on disease modifying factors, and for storage in the Radboudumc biobank for future research (e.g. on biomarkers). Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants will be asked for a visit to the outpatient clinic at the department of neurology. Their medical history will be taken and they will undergo a clinical examination. Several questionnaires can be completed at home through on online system (Castor). Blood samples will be collected in adult patients, a magnetic resonance imaging (MRI) of muscles of both legs (in adults and adolescents) and muscle ultrasound of multiple skeletal muscles will be performed. Spirometry will be performed in a small subset of adult participants. We classify the risk of this study as negligible.

ELIGIBILITY:
Inclusion Criteria:

* All 162 genetically confirmed FSHD patients that participated in the FSHD-FOCUS 2 and 18 genetically conformed pediatric FSHD patient that participated in the FSHD-iFocus study and are informed about the genetic confirmation of FSHD. The 65 newly included patients need to provide genetical confirmation of the disease.

Exclusion Criteria:

* No incapacitated persons will be included in this study. Persons with contra-indications for MRI-scan are excluded for that one procedure, but can be included in the study. Contraindications for MRI-scan include metallic implants (vascular clips, foreign bodies like metallic splinters in the eye, coronary and peripheral artery stents, prosthetic heart valves, pacemakers and ICD's, cochlear implants, breast tissue expanders and some other electronic implants or devices), renal insufficiency, previous allergic reaction to contrast fluids and known claustrophobia.
* Participant in medication trial

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: FSHD patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity to change | 10 years after baseline
  - determine the sensitivity to change of multiple traditional and new clinical outcome measures, patient reported outcome measures and muscle imaging techniques on FSHD
Imaging | 10 years after baseline
  -provide detailed clinical and muscle imaging data on FSHD with a longitudinal follow-up of ten years (T0: baseline FSHD-study T1: five year follow-up or FOCUS-2 study; T2: FOCUS-3 study) to anticipate change in muscle imaging data
Predict disease progression | 10 years after baseline
  - Identification of patterns in disease progression to predict personalized disease trajectories and identify disease modifiers

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided